CLINICAL TRIAL: NCT03318016
Title: Phase I Trial of Arsenic Trioxide With Cyclophosphamide in Patients With Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: Arsenic Trioxide With Cyclophosphamide in Patients With Relapsed/Refractory Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low enrollment, University Scientific Review Committee required study closure.
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 17-0754.cc; NCI-2017-02403 (Other: CTRP)
Record Dates: First submitted 2017-10-18; First posted 2017-10-23 (Actual); Results first posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-02

CONDITIONS: Acute Myeloid Leukemia; Relapsed/Refractory Acute Myeloid Leukemia
Keywords: Arsenic Trioxide; Cyclophosphamide
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: * Cohort -1 (3-6 subjects, if needed): Cyclophosphamide 500 mg/m2
  * Cohort 1 (3-6 subjects): Cyclophosphamide 1000 mg/m2
  * Cohort 2 (3-6 subjects): Cyclophosphamide 2000 mg/m2
  * Cohort 3 (3-6 subjects): Cyclophosphamide 3000 mg/m2
  * Cohort 4 (3 subjects): Cyclophosphamide 4000 mg/m2
  ATO and Cyclophosphamide will be repeated every 28 days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort -1 (Experimental): 3 consecutive days of ATO at a fixed dose of 0.15 mg/kg/d IV followed by Cyclophosphamide on day 4 as a single IV
  Interventions: Drug: Cyclophosphamide 500 MG
- Cohort 1 (Experimental): 3 consecutive days of ATO at a fixed dose of 0.15 mg/kg/d IV followed by Cyclophosphamide on day 4 as a single IV
  Interventions: Drug: Cyclophosphamide 1000 MG
- Cohort 2 (Experimental): 3 consecutive days of ATO at a fixed dose of 0.15 mg/kg/d IV followed by Cyclophosphamide on day 4 as a single IV
  Interventions: Drug: Cyclophosphamide 2000 MG
- Cohort 3 (Experimental): 3 consecutive days of ATO at a fixed dose of 0.15 mg/kg/d IV followed by Cyclophosphamide on day 4 as a single IV
  Interventions: Drug: Cyclophosphamide 3000 MG
- Cohort 4 (Experimental): 3 consecutive days of ATO at a fixed dose of 0.15 mg/kg/d IV followed by Cyclophosphamide on day 4 as a single IV
  Interventions: Drug: Cyclophosphamide 4000 MG

INTERVENTIONS:
Drug: Cyclophosphamide 500 MG — ATO at a fixed dose of 0.15 mg/kg/d IV followed by Cyclophosphamide 500 mg/m2 on day 4 as a single IV dose along with hydration for a maximum of 6 doses
  Other Names: cytophosphane
  Arms: Cohort -1
Drug: Cyclophosphamide 1000 MG — Enrolled subjects will receive 3 consecutive days of ATO at a fixed dose of 0.15 mg/kg/d IV followed by Cyclophosphamide 1000 mg/m2on day 4 as a single IV dose along with Mesna (in subjects receiving ≥1000mg/m2 Cy) and hydration for a maximum of 6 doses
  Other Names: cytophosphane
  Arms: Cohort 1
Drug: Cyclophosphamide 2000 MG — Enrolled subjects will receive 3 consecutive days of ATO at a fixed dose of 0.15 mg/kg/d IV followed by Cyclophosphamide 2000 mg/m2on day 4 as a single IV dose along with Mesna (in subjects receiving ≥1000mg/m2 Cy) and hydration for a maximum of 6 doses
  Other Names: cytophosphane
  Arms: Cohort 2
Drug: Cyclophosphamide 3000 MG — Enrolled subjects will receive 3 consecutive days of ATO at a fixed dose of 0.15 mg/kg/d IV followed by Cyclophosphamide 3000 mg/m2on day 4 as a single IV dose along with Mesna (in subjects receiving ≥1000mg/m2 Cy) and hydration for a maximum of 6 doses
  Other Names: cytophosphane
  Arms: Cohort 3
Drug: Cyclophosphamide 4000 MG — Enrolled subjects will receive 3 consecutive days of ATO at a fixed dose of 0.15 mg/kg/d IV followed by Cyclophosphamide 4000 mg/m2on day 4 as a single IV dose along with Mesna (in subjects receiving ≥1000mg/m2 Cy) and hydration for a maximum of 6 doses
  Other Names: cytophosphane
  Arms: Cohort 4

SUMMARY:
Determine the maximum tolerated dose (MTD) and toxicity profile of the combination of cyclophosphamide and ATO (Arsenic Trioxide) in subjects with relapsed refractory AML.

Determine the efficacy of ATO and cyclophosphamide in this population, as defined by response rate, response duration, event-free survival (EFS) and overall survival (OS).

Determine the number of transplant-eligible subjects who are successfully bridged to stem cell transplantation or donor lymphocyte infusion.

DETAILED DESCRIPTION:
This is an open label phase 1 study of fixed dose ATO (Arsenic Trioxide) and escalating doses of cyclophosphamide using a standard 3+3 dose escalation design. All subjects will be treated with sequential cycles of 3 days of ATO at 0.15 mg/kg/d IV followed by Cyclophosphamide as a single IV dose on day 4 along with mesna at a dose equal to the cyclophosphamide (for doses ≥1000 mg/m2) and hydration for a maximum of 6 cycles. ATO and Cyclophosphamide will be repeated every 28-42 days. Treatment will be given inpatient for the first cycle, with the option of outpatient treatment for subsequent cycles. Subjects may remain on study in the absence of disease progression or unacceptable toxicity for a maximum six cycles. Toxicity assessments will be performed continuously; DLT determination will be made based on adverse events (AEs) that occur during cycle 1 (day 1-28). An expansion cohort of ten subjects at the maximum tolerated dose will occur at the conclusion of dose escalation.

ELIGIBILITY:
Inclusion Criteria:

1. WHO-confirmed AML, other than APL, with no standard treatment options available
2. Age 18 years or older
3. Relapsed or refractory (resistant) disease, as defined by standard criteria

   * Relapsed: Bone marrow blasts ≥5%, reappearance of blasts in the blood, or development of extramedullary disease following achievement of CR/CRi/CRp/MLFS
   * Refractory (resistant): Failure to achieve CR/CRi/MLFS in subjects who survive ≥7 days following completion of initial treatment, with evidence of persistent leukemia by blood and/or bone marrow examination
4. >14 days since any prior therapy for AML excluding hydroxyurea
5. Willing and able to understand and voluntarily sign a written informed consent
6. Able to adhere to the study visit schedule and other protocol requirements
7. Women of childbearing potential must use an acceptable form of birth control for 28 days prior to beginning study treatment, through the duration of study treatment, and for 3 months after discontinuing study treatment.

Exclusion Criteria:

1. New York Heart Association Class III or IV heart failure
2. Unstable angina pectoris
3. Significant uncontrolled cardiac arrhythmias, including ventricular arrhythmias, congenital long QT syndrome, symptomatic atrial fibrillation, symptomatic bradycardia, right bundle branch block plus left anterior hemiblock or bifasicular block
4. QTc >500 ms, uncorrectable by managing electrolytes and medications, using the QTcF formula in Appendix D.
5. Active acute graft vs. host disease ≥ grade 2 or active extensive chronic GVHD
6. Relapse after allogeneic stem cell transplantation prior to post-transplant day 30
7. Active central nervous system (CNS) involvement of leukemia (lumbar puncture not required to rule out CNS involvement if not suspected)
8. Uncontrolled psychiatric illness that would limit compliance with requirements
9. Pregnant or breast feeding females
10. Laboratory abnormalities:

    1. Either creatinine >2.0 mg/dL or creatinine clearance <30 mL/min
    2. Total bilirubin > 3 x institutional upper limit of normal (ULN) (unless documented Gilbert's syndrome)
    3. AST or ALT > 3 x institutional ULN, unless felt to be due to disease involvement
11. Other medical or psychiatric illness or organ dysfunction or laboratory abnormality which, in the opinion of the investigator, would compromise the subject's safety or interfere with data interpretation.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2021-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Pollyea, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort -1: ATO at a fixed dose of 01.15 mg/kg/d IV followed by Cyclophosphamide 500mg/m2 on day 4 as a single IV dose along with hydration for a maximum of 6 doses
- Cohort 1: ATO at a fixed dose of 01.15 mg/kg/d IV followed by Cyclophosphamide 1000 mg/m2 on day 4 as a single IV dose along with Mesna (in subjects receiving > 1000 mg/m2 Cy) and hydration for a maximum of 6 doses
- Cohort 2: ATO at a fixed dose of 01.15 mg/kg/d IV followed by Cyclophosphamide 2000 mg/m2 on day 4 as a single IV dose along with Mesna (in subjects receiving > 1000 mg/m2 Cy) and hydration for a maximum of 6 doses
- Cohort 3: ATO at a fixed dose of 01.15 mg/kg/d IV followed by Cyclophosphamide 3000 mg/m2 on day 4 as a single IV dose along with Mesna (in subjects receiving > 1000 mg/m2 Cy) and hydration for a maximum of 6 doses
- Cohort 4: ATO at a fixed dose of 01.15 mg/kg/d IV followed by Cyclophosphamide 4000 mg/m2 on day 4 as a single IV dose along with Mesna (in subjects receiving > 1000 mg/m2 Cy) and hydration for a maximum of 6 doses
Period: Overall Study
Arm/Group | Cohort -1 | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 0 | 3 | 2 | 0 | 0
Completed | 0 | 3 | 2 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Relapsed/Refractory Acute Myeloid Leukemia
Groups:
- Cohort -1: ATO at a fixed dose of 0.15 mg/kg/d IV followed by Cyclophosphamide 500 mg/m2 on day 4 as a single IV dose along with hydration for a maximum of 6 doses
- Cohort 1: ATO at a fixed dose of 0.15 mg/kg/d IV followed by Cyclophosphamide 1000 mg/m2 on day 4 as a single IV dose along with Mesna (in subjects receiving ≥1000mg/m2 Cy) and hydration for a maximum of 6 doses
- Cohort 2: ATO at a fixed dose of 0.15 mg/kg/d IV followed by Cyclophosphamide 2000 mg/m2 on day 4 as a single IV dose along with Mesna (in subjects receiving ≥1000mg/m2 Cy) and hydration for a maximum of 6 doses
- Cohort 3: ATO at a fixed dose of 0.15 mg/kg/d IV followed by Cyclophosphamide 3000 mg/m2 on day 4 as a single IV dose along with Mesna (in subjects receiving ≥1000mg/m2 Cy) and hydration for a maximum of 6 doses
- Cohort 4: ATO at a fixed dose of 0.15 mg/kg/d IV followed by Cyclophosphamide 4000 mg/m2 on day 4 as a single IV dose along with Mesna (in subjects receiving ≥1000mg/m2 Cy) and hydration for a maximum of 6 doses
- Total: Total of all reporting groups
Arm/Group | Cohort -1 | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total
Number analyzed (Participants) | 0 | 3 | 2 | 0 | 0 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 |  |  | 0
  Between 18 and 65 years | 0 | 0 | 0 |  |  | 0
  >=65 years | 0 | 3 | 2 |  |  | 5
Age, Continuous [Median (Full Range); unit: years] |  | 72 [72 to 82] | 68 [68 to 86] |  |  | 78 [68 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 3 | 0 |  |  | 3
  Male |  | 0 | 2 |  |  | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 0 | 0 |  |  | 0
  Not Hispanic or Latino |  | 3 | 2 |  |  | 5
  Unknown or Not Reported |  | 0 | 0 |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0 |  |  | 0
  Asian |  | 0 | 0 |  |  | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0 |  |  | 0
  Black or African American |  | 0 | 0 |  |  | 0
  White |  | 3 | 2 |  |  | 5
  More than one race |  | 0 | 0 |  |  | 0
  Unknown or Not Reported |  | 0 | 0 |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 3 | 2 |  |  | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Reached Maximally Tolerated Dose (MTD) of Cyclophosphamide and ATO
Description: Number of Participants that were treated in each Cohort in attempt to establish Maximally Tolerated Dose (MTD) of cyclophosphamide with ATO is defined as the highest dose level of 1000 mg/m2. MTD is established when at least 6 participants within a Cohort have responded without toxicity.
  The trial is organized in a standard, phase I, 3+3 design. The first 3 subjects will be assigned to cohort 1. Per standard trial design, if there are 0/3 dose-limiting toxicities (DLT) in this cohort, the next three subjects will be assigned to cohort 2. This will continue until MTD is established.
Time Frame: 26 months
Population: Patients With Relapsed/Refractory Acute Myeloid Leukemia
Measure: Count of Participants; unit: Participants
Groups:
- Cohort -1: Cyclophosphamide: ATO at a fixed dose of 0.15 mg/kg/d IV followed by Cyclophosphamide 500 mg/m2 on day 4 as a single IV dose along with hydration for a maximum of 6 doses.
- Cohort 1: Cyclophosphamide: ATO at a fixed dose of 0.15 mg/kg/d IV followed by Cyclophosphamide 1000 mg/m2 on day 4 as a single IV dose along with Mesna (in subjects receiving >1000mg/m2 Cy) and hydration for a maximum of 6 doses
- Cohort 2: Cyclophosphamide: ATO at a fixed dose of 0.15 mg/kg/d IV followed by Cyclophosphamide 2000 mg/m2 on day 4 as a single IV dose along with Mesna (in subjects receiving >1000mg/m2 Cy) and hydration for a maximum of 6 doses
- Cohort 3: Cyclophosphamide: ATO at a fixed dose of 0.15 mg/kg/d IV followed by Cyclophosphamide 3000 mg/m2 on day 4 as a single IV dose along with Mesna (in subjects receiving >1000mg/m2 Cy) and hydration for a maximum of 6 doses
- Cohort 4: Cyclophosphamide: ATO at a fixed dose of 0.15 mg/kg/d IV followed by Cyclophosphamide 4000 mg/m2 on day 4 as a single IV dose along with Mesna (in subjects receiving >1000mg/m2 Cy) and hydration for a maximum of 6 doses
Arm/Group | Cohort -1 | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 0 | 3 | 2 | 0 | 0
Participants | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Overall Response Rate (ORR) Using ATO and Cyclophosphamide
Description: ORR defined by complete remission/complete remission with incomplete recovery of blood counts (CR/CRi), morphologic leukemia free state (MLFS) and partial responses (PR)
Time Frame: 26 months
Population: Subjects provided both ATO and Cyclophosphamide
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort -1 | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 0 | 3 | 2 | 0 | 0
Participants |  | 3 | 2 |  |

ADVERSE EVENTS:
Time Frame: 26 months
Description: Some cohorts did not accrue any subjects. Therefor, the number of Serious Adverse Events, All-Cause Mortality and Other Adverse Events is zero.
Arm/Group | Cohort -1 | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/3 | 0/2 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 1/3 | 0/2 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 3/3 | 2/2 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort -1 (N=0) | Cohort 1 (N=3) | Cohort 2 (N=2) | Cohort 3 (N=0) | Cohort 4 (N=0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | NA | 1 (1) | NA | NA | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | NA (0) | 1 (1) | NA | NA | NA
Chest Pain (Respiratory, thoracic and mediastinal disorders) | NA | 1 (1) | NA | NA | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort -1 (N=0) | Cohort 1 (N=3) | Cohort 2 (N=2) | Cohort 3 (N=0) | Cohort 4 (N=0)
Activity Change (General disorders) | NA | 1 (1) | 0 (0) | NA | NA
Pain (Musculoskeletal and connective tissue disorders) | NA | 1 (1) | 1 (1) | NA | NA
Acute Kidney Injury (Renal and urinary disorders) | NA | 1 (1) | 0 (0) | NA | NA
Anemia (Blood and lymphatic system disorders) | NA | 0 (0) | 1 (1) | NA | NA
Anorexia (General disorders) | NA | 1 (1) | 1 (1) | NA | NA
Anxiety (Psychiatric disorders) | NA | 1 (1) | 0 (0) | NA | NA
Appetite Change (General disorders) | NA | 1 (1) | 0 (0) | NA | NA
Chest pain (Respiratory, thoracic and mediastinal disorders) | NA | 1 (1) | 0 (0) | NA | NA
chills (Respiratory, thoracic and mediastinal disorders) | NA | 1 (1) | 0 (0) | NA | NA — Related to pneumonia diagnosis
Cough (Respiratory, thoracic and mediastinal disorders) | NA | 1 (2) | 1 (1) | NA | NA
Dehydration (Metabolism and nutrition disorders) | NA | 0 (0) | 1 (1) | NA | NA
Depression (Psychiatric disorders) | NA | 0 (0) | 1 (1) | NA | NA
Dyspnea (Respiratory, thoracic and mediastinal disorders) | NA | 1 (1) | 0 (0) | NA | NA
Edema (Blood and lymphatic system disorders) | NA | 2 (2) | 1 (1) | NA | NA
Creatinine Increase (Renal and urinary disorders) | NA | 0 (0) | 1 (1) | NA | NA
epistaxis (Skin and subcutaneous tissue disorders) | NA | 2 (2) | 0 (0) | NA | NA
Fatigue (General disorders) | NA | 1 (1) | 0 (0) | NA | NA
Fever (General disorders) | NA | 2 (2) | 0 (0) | NA | NA
Alopecia (Skin and subcutaneous tissue disorders) | NA | 1 (1) | 0 (0) | NA | NA
Hypocalcemia (Blood and lymphatic system disorders) | NA | 1 (1) | 1 (1) | NA | NA
Hypophosphatemia (Blood and lymphatic system disorders) | NA | 1 (1) | 1 (1) | NA | NA
Hypotension (Blood and lymphatic system disorders) | NA | 0 (0) | 1 (1) | NA | NA
Hyponatremia (Blood and lymphatic system disorders) | NA | 1 (1) | 0 (0) | NA | NA
Constipation (Metabolism and nutrition disorders) | NA | 0 (0) | 1 (1) | NA | NA
Hypomagnesia (Blood and lymphatic system disorders) | NA | 1 (1) | 0 (0) | NA | NA
Sensory neuropathy (Nervous system disorders) | NA | 0 (0) | 1 (1) | NA | NA
Lip ulcer (General disorders) | NA | 1 (1) | 0 (0) | NA | NA
Myalgia (Musculoskeletal and connective tissue disorders) | NA | 1 (1) | 0 (0) | NA | NA
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | NA | 1 (1) | 0 (0) | NA | NA
Pallor (Blood and lymphatic system disorders) | NA | 1 (1) | 0 (0) | NA | NA
prolonged QTc (Cardiac disorders) | NA | 1 (1) | 0 (0) | NA | NA
rash (Skin and subcutaneous tissue disorders) | NA | 1 (1) | 0 (0) | NA | NA
Skin infection (Skin and subcutaneous tissue disorders) | NA | 1 (1) | 0 (0) | NA | NA
skin tear (Skin and subcutaneous tissue disorders) | NA | 1 (1) | 0 (0) | NA | NA
tarry stool (Metabolism and nutrition disorders) | NA | 1 (1) | 0 (0) | NA | NA
throat irritation (General disorders) | NA | 1 (1) | 0 (0) | NA | NA
thrombophlebitis (Blood and lymphatic system disorders) | NA | 1 (1) | 0 (0) | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-10-16): https://cdn.clinicaltrials.gov/large-docs/16/NCT03318016/Prot_SAP_ICF_000.pdf